CLINICAL TRIAL: NCT02172027
Title: Novel Immunomagnetic Detection of Cancer Cells in Pleural Effusion in Lung Cancer Patients as Additional Staging and Prognostic Tool
Brief Title: Immunomagnetic Detection of Cancer Cells in Pleural Effusion in Lung Cancer Patients as Additional Staging and Prognostic Tool
Status: Withdrawn | Type: Observational
Why Stopped: Technical problems with the device
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ImmunoMag-Det LC 00432014
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2014-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung Cancer, Pleural effusion
  Interventions: Device: Immunomagnetic Detection

INTERVENTIONS:
Device: Immunomagnetic Detection — Analysis of pleural effusion through immunomagnetic detection device.
  Other Names: BioCep

SUMMARY:
Pleural effusion in lung cancer patients is one of the symptoms of metastatic disease that is inoperable and cannot be treated. Identification of cancer cells in the pleural effusion of lung cancer patients is a cytological test and serves as an initial diagnosis. These cells can then be used to prepare a cell block for staining and further tests.

In some research despite clinical suspicions, the cytological diagnosis is negative, due to the specimen containing too few cells or damage to the cells whilst the specimen is processed. A new method of identifying rare cells in a fluid is by immunomagnetic separation. Using this method, an antigen binds to proteins in the cell wall that are unique to tumor cells. When the fluid is passed through a magnetic field, separation occurs of the cells with the magnetic tags from the remainder of the cells. The separated cells can then be stained or cultured.

The currently approved method of immunomagnetic detection has been approved for clinical use in patients with breast cancer, cancer of the intestines and prostate cancer. An Israeli Biotech company has developed an advanced technology that allows identification of a larger number of cells without causing morphological damage to the cells.

The purpose of the current study is to examine the technique of immunomagnetic separation in pleural effusion of lung cancer patients in comparison to the cytological tests. In the future it is hoped that a larger number of patient samples will be included and further characterization of the cells will be possible to be compared to the clinical and cytological characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Lung Cancer Patients in the Lung Department or Oncology Department with spread to the pleural cavity.

Exclusion Criteria:

* Under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients with pleural effusion at the Meir Medical Center Oncology Department or Lung Department.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To compare the method of Immunomagnetic detection to the current cytological test. | The samples will analyzed within a year
  The sample will be sent in parallel for cytological testing and immunomagnetic separation. By comparing the percentage of positive cells identified by the two methods of analysis, it can be determined whether immunomagnetic separation is an efficient method of identifying cancerous cells.

SECONDARY OUTCOMES:
The sensitivity of the technique of immunomagnetic separation compared to existing cytological techniques. | Within two years
  The sensitivity of the new technique of immunomagnetic separation will be assessed through analysis of the percentage of positive cells identified compared to the gold standard of cytological techniques.